CLINICAL TRIAL: NCT02897882
Title: Acute and Chronic Pain in Lung Transplantation: Prevalence, Associated Factors, Medical Care
Brief Title: Acute and Chronic Pain in Lung Transplantation: Prevalence, Associated Factors, Taken Care
Acronym: MUCODOULEUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2009/58; 2009-A01353-54 (Other: ANSM)
Record Dates: First submitted 2016-08-31; First posted 2016-09-13 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung transplant (Experimental): Pain evaluation
  Interventions: Other: Lung transplant

INTERVENTIONS:
Other: Lung transplant — Pain evaluation

SUMMARY:
The objective of this project is to estimate the frequency and the characters of the chronic pains by a follow-up which begins during the registration on the waiting list of transplant and which ends at the end of the third year following the lung transplantation. It is a forward-looking study of prevalence entering within the framework of the common care. After lung transplant, pain will be evaluate with questionnaires every day during the hospitalisation, and then after 1 month, 3 months, 6 months, 1 year, 2 years and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients benefiting from a lung transplant
* Patients on a list for a lung transplant from may 2010

Exclusion Criteria:

* Patients refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Chronic pain measured by a digital scale | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, PhD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No